CLINICAL TRIAL: NCT02475005
Title: An Intervention to Improve Adolescent Headache Self-management
Acronym: TH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stephen F Butler, PhD (Industry)
Responsible Party: Sponsor-Investigator, Stephen F Butler, PhD, Senior VP/Chief Science Officer, Inflexxion, Inc.
Organization: Inflexxion, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2R44HD066920-03A1 (NIH)
Record Dates: First submitted 2015-06-12; First posted 2015-06-18 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Pain; Headache
Keywords: self management app; headache; adolescent
MeSH Terms: conditions — Pain; Headache

ARMS (2):
- Mobile self management app on smartphone (Experimental): Mobile self management app on smartphone
  Interventions: Behavioral: pain self management app on smartphone
- Treatment as usual (No Intervention): Treatment as usual (control group)

INTERVENTIONS:
Behavioral: pain self management app on smartphone
  Arms: Mobile self management app on smartphone

SUMMARY:
The purpose of this study is to test the efficacy of a new app to help adolescents with chronic or reoccurring headaches self manage pain.

DETAILED DESCRIPTION:
Headaches dramatically affect adolescents' overall functioning and quality of life. We have developed a highly engaging mobile-based program that will help adolescents to make connections between behaviors and symptoms, and to ultimately improve functioning and quality of life. The mobile-based program will provide a state of the art pain tracker, a variety of coping strategies, and information about self-management of symptoms. This app will offer a maximally engaging way to help adolescents track their pain, make connections between lifestyle and pain, and learn key self-management skills.

The study involves the participant being randomized into either the experimental group, where he/she will be using this mobile application to track their headache symptoms, or the control group, where he/she will receive headache treatment as usual; the control group will not be using an app for this study. The intervention will last for two months.

Participants will be assessed at baseline, at 2-months post baseline, at 3-months post baseline, and at 6-months post baseline. All participants will be asked to complete online questionnaires about their headaches. We plan to enroll 144 adolescent participants with headaches, as well as one caregiver (meaning a parent/guardian) for each adolescent.

ELIGIBILITY:
[The above age limits are specific to adolescent participants.]

Inclusion Criteria - Adolescents

* Between ages 13 and 17 (inclusive)
* Able to read and speak English
* Has recurring headaches that are not related to another medical condition
* iPhone user with access to an iPhone [4/4S or later] for use during the intervention period

Exclusion Criteria - Adolescents

* Secondary headache or seizure disorder. Examples include: increased intracranial pressure, hydrocephalus, traumatic brain injury, benign or cancerous brain
* Cognitive impairment or psychiatric condition that would interfere with ability to use the mobile application or complete the assessments

Inclusion Criteria - Caregivers

Parent or guardian of an adolescent who meets the above eligibility criteria for adolescent participants

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2014-09-20 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Change in pain coping at 2 months, 3 months, and 6 months post-baseline | 2 months, 3 months, 6 months
  Measured by Pain Coping Questionnaire (PCQ) - Reid et al., 1998
Change in headache intensity at 2 months, 3 months, and 6 months post-baseline | 2 months, 3 months, 6 months
  "In the past 7 days, how would you rate your headache pain on average..." from 0-no pain to 10-worst possible pain
Change in headache frequency at 2 months, 3 months, and 6 months post-baseline | 2 months, 3 months, 6 months
  On how many days during the past 30 days have you had a headache? How many days in the past 30 were you completely headache free?"
Change in quality of life at 2 months, 3 months, and 6 months post-baseline | 2 months, 3 months, 6 months
  Measured by PedMIDAS - Hershey et al., 2001

SECONDARY OUTCOMES:
Change in pain self-efficacy at 2 months, 3 months, and 6 months post-baseline | 2 months, 3 months, 6 months
  Measured by Pain Self-Efficacy Scale - Burch, Tsao, et al., 2006
Change in school absenteeism at 2 months, 3 months, and 6 months post-baseline | 2 months, 3 months, 6 months
  Ask caregivers: "How many full school days did your child miss in the past 30 days due to headaches?"
Change in physical and psychosocial functioning at at 2 months, 3 months, and 6 months post-baseline | 2 months, 3 months, 6 months
  Measured by parent report version of the PedsQL 4.0 (Varni et al., 1999)
Change in health care utilization at 2 months, 3 months, and 6 months post-baseline | 2 months, 3 months, 6 months
  Measured by asking caregiver to report information such as the following:
  * How many days in the past 30 days did his/her child see a healthcare provider for his/her headaches?
  * What types of treatment (including medications) has his/her child received for headaches in the past 30 days?

CONTACTS AND LOCATIONS:
Locations (1):
- Inflexxion, Newton, Massachusetts, United States